CLINICAL TRIAL: NCT07187713
Title: ACE Reno, Effect of Pico Cell Matrix on Patients With Micro-albuminuria, Proteinuria or CKD (of Any Degree) Due to Diabetes Mellitus, Autoimmune, Miscellaneous Aetiology
Brief Title: ACE Reno, Pico Cell Matrix and Its Effect on eGFR in Chronic Kidney Diseases
Acronym: ACE Reno
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ace Cells Lab Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACE_Reno
Record Dates: First submitted 2025-09-07; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Hypertensive Nephropathy; Auto Immune Disorders; Chronic Kidney Disease; Chronc Kidney Disease Stage 5; Chronic Kidney Disease (Stage 3-4); Chronic Kidney Disease (Stages 4 and 5); Microalbuminuria; Diabetic Nephropathies
Keywords: chronic kidney disease; ckd; nephropathy
MeSH Terms: conditions — Hypertensive Nephropathy; Renal Insufficiency, Chronic; Diabetic Nephropathies; Kidney Diseases

STUDY DESIGN:
Intervention Model Description: 1 ml sublingually 4 times a day for 12 weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 1 ml sublingual 4 times daily for 12 weeks (Experimental): Participants will receive ACE Reno, a standardized oral transmucosal solution containing low-molecular-weight bioactive peptides and amino acids.
  The formulation is designed to engage antifibrotic (BMP-7-like, HGF-like, Klotho-like) and vasodilatory/natriuretic peptide-like pathways relevant to glomerular and tubulointerstitial function.
  No genetic material is present; formulation is peptide-based only.
  Interventions: Drug: ACE Reno

INTERVENTIONS:
Drug: ACE Reno — 1 ml sublingual 4 times daily for 12 weeks

SUMMARY:
This study investigates the safety and efficacy of ACE Reno, an oral transmucosal solution containing standardized bioactive peptides and amino acids, in patients with nephropathy of various etiologies and stages. The trial evaluates whether 12 weeks of ACE Reno (1 mL sublingually four times daily) reduces albuminuria/proteinuria and stabilizes kidney function in participants with nephropathy due to diabetes, hypertension, autoimmune disease, reflux/UTI, chronic glomerulonephritis, unknown etiology, pre-dialysis CKD, or post-transplant proteinuria.

Nephropathy remains a global health burden, with ~9-10% of the population affected by chronic kidney disease (CKD), equating to >750 million individuals worldwide. The socioeconomic costs are substantial: in England CKD costs ~£7 billion annually, projected to rise to ~£14 billion by 2033; in Malaysia, prevalence rose from 9% to 15.5% within 7 years; in Egypt, CKD imposes heavy familial and financial burdens, especially for pediatric patients; in Turkey, CKD is among the top causes of disability, linked to the rising tide of diabetes, obesity, and hypertension.

ACE Reno is designed to address multiple drivers of CKD progression - glomerulosclerosis, fibrosis, endothelial dysfunction, and maladaptive RAAS/aldosterone signaling - through its peptide components that mimic antifibrotic (BMP-7, HGF, Klotho-like) and vasodilatory/cGMP-mediated (natriuretic peptide-like) pathways.

DETAILED DESCRIPTION:
Study Objectives

Primary Objective:

To evaluate the effect of ACE Reno on urinary albumin-to-creatinine ratio (ACR) after 12 weeks of treatment in patients with nephropathy of diverse etiologies.

Secondary Objectives:

To assess the effect of ACE Reno on estimated glomerular filtration rate (eGFR) slope.

To evaluate changes in proteinuria, blood pressure, and patient-reported outcomes.

To assess safety and tolerability.

Exploratory Objectives:

To explore biomarker changes (e.g., TGF-β, cGMP, NGAL, KIM-1). To assess durability of response up to 6 months in responders. Investigational Product (IP) ACE Reno is a sublingual solution (1 mL four times daily for 12 weeks) containing a standardized panel of low-molecular-weight bioactive peptides and amino acids.

Key peptide domains include:

BMP-7-like sequences countering TGF-β-driven fibrosis. HGF-like fragments supporting epithelial repair. Klotho-like motifs antagonizing profibrotic pathways and RAAS/Wnt activity. Natriuretic-peptide-like domains enhancing cGMP signaling, with anti-fibrotic, vasodilatory, and endothelial-protective effects.

No genetic material is present; formulation is peptide-based only. Study Design Type: Prospective, multicenter, interventional, open-label. Model: Single-arm with within-patient comparisons. Duration: 12 weeks treatment + 4 weeks post-treatment safety follow-up. Visits: Screening, Baseline (Day 0), Week 4, Week 8, Week 12, and Week 16 safety call.

Participants

Inclusion:

Adults (≥18 years) with nephropathy of any degree (microalbuminuria, overt proteinuria, CKD stages 1-5 not on dialysis, or post-transplant with proteinuria). Stable background therapy with ACEi/ARB, SGLT2i, or MRA allowed.

Exclusion:

Dialysis at baseline. Recent kidney transplant (<12 months). Uncontrolled acute infection or unstable autoimmune disease. Pregnancy or lactation. Known hypersensitivity to study components. Categories (Strata: 17 Subgroups) Diabetic nephropathy - microalbuminuria Diabetic nephropathy - macroalbuminuria Diabetic nephropathy - CKD Stage 3 Diabetic nephropathy - CKD Stage 4-5 (non-dialysis) Hypertensive nephropathy - microalbuminuria Hypertensive nephropathy - proteinuric CKD Hypertensive nephropathy - advanced CKD (3-5) Autoimmune nephropathy - Class II-III Autoimmune nephropathy - Class IV-V Reflux nephropathy - mild/moderate scarring Reflux nephropathy - severe scarring Chronic glomerulonephritis - nephrotic range proteinuria Chronic glomerulonephritis - CKD <60 mL/min/1.73m² CKD of unknown etiology - Stage 1-2 CKD of unknown etiology - Stage 3-4 ESRD pre-dialysis (eGFR <15) Post-transplant CKD with proteinuria Sample Size and Rationale

Primary endpoint powering (paired design):

Detect 30% reduction in ACR (δ = ln(0.70) = -0.357), assuming σ = 0.8, r = 0.6 → ~32 analyzable patients needed.

Planned enrollment (pooled cohort, with 17 categories):

~182 analyzable patients (~214 enrolled allowing for 15% attrition). Each category will include a minimum of 8-12 patients (more for common etiologies such as diabetic proteinuria).

Total enrollment stratified by prevalence across categories. Endpoints

Primary Endpoint:

Change in urinary ACR from baseline to Week 12 (log-transformed).

Secondary Endpoints:

Change in eGFR slope. Change in 24-h proteinuria (selected patients). Blood pressure change. Patient-reported outcomes (KDQOL-36, EQ-5D). Safety (hyperkalemia, creatinine rise, liver tests, hematology).

Exploratory Endpoints:

Biomarker profiles (TGF-β, cGMP, NGAL, KIM-1). Hospitalization rate. Extended follow-up outcomes at 6 months. Follow-Up Plan

Monthly Visits (Week 4, 8, 12):

Clinical: BP, vitals, weight, adherence. Labs: creatinine/eGFR, electrolytes, liver panel, CBC, urine ACR. Safety: hyperkalemia, creatinine rise. PROs brief (fatigue, QoL).

Final (Week 12):

Primary endpoint assessment (duplicate ACR). PROs full set. Investigator global assessment.

Safety Call (Week 16):

AE/SAE resolution, concomitant therapy updates. Statistical Analysis Primary analysis: Paired t-test and mixed model for repeated measures (MMRM) on log(ACR).

Secondary: eGFR slope via linear mixed model, BP change via ANCOVA, responder rate (≥30% reduction in ACR).

Subgroups: Category-by-time interaction analysis; forest plots for effect estimates.

Multiplicity: Subgroup effects exploratory; overall primary endpoint tested at α=0.05.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years) with nephropathy of any degree (microalbuminuria, overt proteinuria, CKD stages 1-5 not on dialysis, or post-transplant with proteinuria). Stable background therapy with ACEi/ARB, SGLT2i, or MRA allowed.

Exclusion Criteria:

* Recent kidney transplant (<12 months). Uncontrolled acute infection or unstable autoimmune disease. Pregnancy or lactation. Known hypersensitivity to study components.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-09-20 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Urinary Albumin-to-Creatinine Ratio (ACR) | 12 weeks
  Percent change in log-transformed urinary ACR measured from first-morning urine samples. The primary analysis compares baseline to Week 12 values

SECONDARY OUTCOMES:
Change in Estimated Glomerular Filtration Rate (eGFR) slope | Baseline, Week 4, Week 8, Week 12
  eGFR calculated from serum creatinine using CKD-EPI; slope analyzed via linear mixed model.
Change in 24-hour Proteinuria | Baseline to Week 12 (subset of participants with baseline nephrotic-range proteinuria)
  Absolute and percent change in 24-hour urinary protein excretion.
Change in Blood Pressure | Baseline, Week 4, Week 8, Week 12
  tp adjust BP : systolic <=140 Diastolic >100 up to 60 mmHg
Safety and Tolerability | Throughout treatment and up to Week 16 follow-up
  measure 'Full blood count before and after 16 weeks
Safety and Tolerability | Throughout treatment and up to Week 16 follow-up
  measure ALT before and after 16 weeks
Safety and Tolerability | Throughout treatment and up to Week 16 follow-up
  measure 'AST before and after 16 weeks
Safety and Tolerability | Throughout treatment and up to Week 16 follow-up
  measure Bilirubin before and after 16 weeks
Safety and Tolerability | Throughout treatment and up to Week 16 follow-up
  measure 'Urea before and after 16 weeks
Safety and Tolerability | Throughout treatment and up to Week 16 follow-up
  measure 'Creatinine before and after 16 weeks

OTHER OUTCOMES:
Hospitalization Events | Baseline to Week 16
  Number of hospitalizations related to renal or cardiovascular complications.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. Mohammed Yasser Sayyed Saif, PhD, Principal Investigator — Beni Suef Univeristy; Dr. Alaa Abdelkarim M Fouad, MRCPUK SEC, Principal Investigator — British Centre for Regenerative medicine BCRMED
Locations (1):
- British Centre For Regenerative medicine BCRMED Global, Giza, GZ, Egypt

IPD SHARING:
Plan to Share IPD: No